CLINICAL TRIAL: NCT05085171
Title: A Community-based Phase III, Cluster Randomized Trial of Point-of-care CD4 Testing and Enhanced Screening and Prophylaxis in Advanced HIV Disease
Brief Title: An Enhanced Package of Care to Reduce Reduce Mortality in Advanced HIV Disease
Acronym: ENCORE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: IDIREC REF 007/2021
Record Dates: First submitted 2021-10-08; First posted 2021-10-20 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: The Study Will Focus on Assessing the Survival Benefit on an Enhanced Package of Care for Patients With Advanced HIV Disease

STUDY DESIGN:
Intervention Model Description: A community randomised controlled trial of 24 clinics,12 in the intervention arm and 12 in standard of care arm. Two levels of randomization planned
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention(Enhanced package of care) Arm (Experimental): The patients with advanced HIV disease that receive HIV care at the intervention clinics will receive the enhanced intervention package which will include: point of care CD4 testing with visitect, screening for TB and cryptococcal meningitis using Fujifilm LAM and semiquantitative crAg LFA respectively and pre-emptive treatment with isoniazid and rifapentine for one month. Those with a high crAg titers will receive treatment for CNS cryptococcal disease.
  Interventions: Other: Enhanced care package
- Standard of care Arm (No Intervention): The patients with advanced HIV disease that receive HIV care at the standard of care clinics will receive the usual routine HIV care as per the Uganda national guidelines. That is CD4 testing with flowcytometry or other CD4 testing modalities available, screening for TB and cryptococcal meningitis using Alere LAM and crAg LFA respectively and pre-emptive treatment with isoniazid and rifapentine for 3-6 month. Treatment of all asymptomatic crAG positives with fluconazole as per guidelines.

INTERVENTIONS:
Other: Enhanced care package — The intervention is an improved package of care for patients with advanced HIV disease with point of care CD4 testing, more sensitive screening tests for opportunistic infections and more intensive pre-emptive treatment for opportunistic infections
  Arms: intervention(Enhanced package of care) Arm

SUMMARY:
A community-based Phase III, cluster randomized trial that seeks to determine the 24 week survival with retention in care of point of care CD4 testing with visitect and an enhanced package of screening and prophylaxis for opportunistic infections among patients with advanced HIV disease.

DETAILED DESCRIPTION:
The study will be carried out in a population of HIV-infected adults with advanced HIV disease (CD4 <200 cells/µL) in Uganda. It will be a Randomized controlled trial, Phase III in Uganda over a duration of 5 years assessing 24 weeks survival with retention in care. @4 clinic will be randomized to either receive the enhanced package or standard of care.

Description of Intervention Arm

1. Point-of-care CD4 testing via Visitect (point of care semi Quantitaive CD4 LFA) lateral flow assay (LFA)
2. Enhanced package of opportunistic infection screening and prophylaxis for CD4<200, including:

   * FujiFilm SILVAMP TB LAM (FujiLAM)
   * Isoniazid (INH) + rifapentine: 1 month of therapy for latent TB(Tuberculosis) infection
   * Cryptococcal Antigen semi-quantitative (CrAg-SQ) LFA (Immy)
   * Treatment for disseminated CNS cryptococcal infection if high blood CrAg titer (>3+ CrAg SQ)

Description of Standard of Care Arm

1. CD4 testing by flow cytometry
2. WHO recommended package of OI screening and prophylaxis, including:

   * Urine TB LAM
   * INH ( isoniazid 6 months)
   * CrAg LFA
   * Fluconazole for asymptomatic CrAg+ o 800mg daily x 2 weeks, then 400mg daily x 8 weeks, then 200mg daily.

Problem statement: Current lab-based CD4 testing results in a delay to either start ART(Antiretroviral therapy) or a delay in screening persons with low CD4s for OIs. At present, prioritization has been on ART initiation without systematic OI screening. Those with subclinical OIs started on ART unmask their OIs, with hospitalization / deaths for OIs such as cryptococcosis and TB.

We hypothesize that with point of care CD4 testing, same-day OI screening can occur, yet not interrupt prompt ART initiation for those at low risk (FujiLAM and CrAg-SQ negative) of unmasking immune reconstitution syndrome.

We hypothesize that point-of-care CD4 testing will improve 6-month survival by reducing lag time in CD4 results, thereby facilitating ART initiation, retention-in-care, and OI screening and prophylaxis.

We hypothesize that enhanced screening with the point-of-care FujiLAM, CrAg-SQ LFA, with enhanced prophylaxis for TB (1 month of INH and rifapentine) and with treatment for disseminated CNS cryptococcal infection in those CrAg+ with high titers (>3+) will improve 6-month survival compared to current WHO-recommended standard practice in persons with advanced HIV disease.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* CD4<200 cells/µL
* Ability and willingness to give informed consent for the enhanced package of care arm.

Exclusion Criteria:

* Known virologic suppression (viral load <1000 copies/mL) within prior 3 months
* Cannot or unlikely to attend regular clinic visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
24-week survival with retention in care | 24 weeks
  Comparison will be made between study arms of those who receive POC CD4 testing vs. those who receive standard flow cytometry, and those who receive the enhanced package of OI screening and prophylaxis, vs. those who receive the current WHO standard.

SECONDARY OUTCOMES:
Evaluate sensitivity and specificity of the different TB point of care tests. | 24 weeks
  After a positive FujiFilm TB LAM test, incidence of Xpert-positive or culture positive TB, and clinical outcomes to distinguish between false positive vs. true positive urine tests
Incidence of OIs and associated hospitalization and mortality | Six months
  Incidence of active TB within 6 months, Incidence of cryptococcal meningitis and associated mortality.
Tolerability and adherence to prophylaxis regimen and associated grade 3 to 5 adverse events | 24 weeks
  percentage completion of regimen and proportions that get grade 3 and above AEs.

CONTACTS AND LOCATIONS:
Locations (1):
- kisugu health center IV, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No
Aggregated patient data will be summarized and disseminated.